CLINICAL TRIAL: NCT02645695
Title: Can High Frequency Chest Wall Oscillation Accelerate the Discharged of Intubated Intensive Care Patients?
Brief Title: What is the Effective Pulmonary Physiotherapy Method in Critically Care Patients?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ILKE KUPELI (Other)
Responsible Party: Sponsor-Investigator, ILKE KUPELI, head of Anesthesiology and Reanimation, Erzincan University
Organization: Erzincan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: erzincan university
Record Dates: First submitted 2015-12-30; First posted 2016-01-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Atelectasis
Keywords: Pulmonary Rehabilitation; Chest Physiotherapy; High Frequency Chest Wall Oscillation
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- routine pulmonary rehabilitation (Active Comparator): routine pulmonary rehabilitation consisted of position giving technique
  Interventions: Device: routine pulmonary rehabilitation; Device: chest wall vibration technique
- chest wall vibration technique (Active Comparator): chest wall vibration technique in addition to the routine pulmonary rehabilitation method for 72 hours.
  Interventions: Device: routine pulmonary rehabilitation; Device: chest wall vibration technique

INTERVENTIONS:
Device: routine pulmonary rehabilitation — received routine pulmonary rehabilitation consisted of position giving technique (left lateral, supine, right lateral), chest wall percussion, postural drainage and airway aspiration at every 3 hours.
Device: chest wall vibration technique — administered chest wall vibration technique in addition to the routine pulmonary rehabilitation method for 72 hours. Chest vibration method was applied with 7-10 hz frequency given by a ped wrapped around the thorax and pulmonary rehabilitation with 3 mmHg pressure four times a day with 15-minute periods (TheVest® Model 205).

SUMMARY:
Effects of the high frequent chest wall oscillation technique applied on the patients who were intubated in intensive care unit were investigated.

A total of 30 patients who were intubated and under the mechanical ventilator supplied, were included in the study. While the control group (n=15) received routine pulmonary rehabilitation technique, the study group (n=15) was administered high frequency chest wall oscillation for 72 hours as 4 times of 15-minute intervals, in addition to the pulmonary rehabilitation technique. Patients 'APACHE-II scores, dry sputum weight, Lung Collapse Index and blood gas values were measured at the hours 24th, 48th and 72nd, and endotracheal aspirate culture was studied at initial and 72nd. In addition, patient outcomes were evaluated at the end of the first week.

ELIGIBILITY:
Inclusion Criteria:

* aged over 18 years
* Patients with more than three days intubated, in critical care unit of Mengücekgazi Training and Research Hospital

Exclusion Criteria:

* Patients with rib fracture
* acute hemorrhage
* unstable intracranial pressure
* existence of chest drainage tube and those have history of spinal surgery,
* skin infection in the back and chest area and subcutaneous emphysema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
change from baseline of Lung Collapse Index (LCI) values were recorded by listening both the lungs and scoring between 0 and 4 (0: normal expansion, 1: single lobe collapse, 2: 2 lobe collapse, 3: multiple lobe collapse) at six month | six month

SECONDARY OUTCOMES:
weight of the dry sputum after six month | six month

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Esguerra-Gonzalez A, Ilagan-Honorio M, Fraschilla S, Kehoe P, Lee AJ, Marcarian T, Mayol-Ngo K, Miller PS, Onga J, Rodman B, Ross D, Sommer S, Takayanagi S, Toyama J, Villamor F, Weigt SS, Gawlinski A. CNE article: pain after lung transplant: high-frequency chest wall oscillation vs chest physiotherapy. Am J Crit Care. 2013 Mar;22(2):115-24. doi: 10.4037/ajcc2013869. PMID 23455861
- [Background] Massard G, Wihlm JM. Postoperative atelectasis. Chest Surg Clin N Am. 1998 Aug;8(3):503-28, viii. PMID 9742334
- [Background] Manzano RM, Carvalho CR, Saraiva-Romanholo BM, Vieira JE. Chest physiotherapy during immediate postoperative period among patients undergoing upper abdominal surgery: randomized clinical trial. Sao Paulo Med J. 2008 Sep;126(5):269-73. doi: 10.1590/s1516-31802008000500005. PMID 19099160
- [Result] Ntoumenopoulos G, Presneill JJ, McElholum M, Cade JF. Chest physiotherapy for the prevention of ventilator-associated pneumonia. Intensive Care Med. 2002 Jul;28(7):850-6. doi: 10.1007/s00134-002-1342-2. Epub 2002 May 24. PMID 12122521
- [Result] Ciesla ND. Chest physical therapy for patients in the intensive care unit. Phys Ther. 1996 Jun;76(6):609-25. doi: 10.1093/ptj/76.6.609. PMID 8650276
- [Result] Oermann CM, Swank PR, Sockrider MM. Validation of an instrument measuring patient satisfaction with chest physiotherapy techniques in cystic fibrosis. Chest. 2000 Jul;118(1):92-7. doi: 10.1378/chest.118.1.92. PMID 10893365
- [Result] Warwick WJ, Wielinski CL, Hansen LG. Comparison of expectorated sputum after manual chest physical therapy and high-frequency chest compression. Biomed Instrum Technol. 2004 Nov-Dec;38(6):470-5. doi: 10.2345/0899-8205(2004)38[470:COESAM]2.0.CO;2. PMID 15635998
- [Result] Hansen LG, Warwick WJ, Hansen KL. Mucus transport mechanisms in relation to the effect of high frequency chest compression (HFCC) on mucus clearance. Pediatr Pulmonol. 1994 Feb;17(2):113-8. doi: 10.1002/ppul.1950170207. PMID 8165037
- [Result] Gross D, Zidulka A, O'Brien C, Wight D, Fraser R, Rosenthal L, King M. Peripheral mucociliary clearance with high-frequency chest wall compression. J Appl Physiol (1985). 1985 Apr;58(4):1157-63. doi: 10.1152/jappl.1985.58.4.1157. PMID 3988672
- [Result] Langenderfer B. Alternatives to percussion and postural drainage. A review of mucus clearance therapies: percussion and postural drainage, autogenic drainage, positive expiratory pressure, flutter valve, intrapulmonary percussive ventilation, and high-frequency chest compression with the ThAIRapy Vest. J Cardiopulm Rehabil. 1998 Jul-Aug;18(4):283-9. doi: 10.1097/00008483-199807000-00005. PMID 9702607
- [Result] Chen YC, Wu LF, Mu PF, Lin LH, Chou SS, Shie HG. Using chest vibration nursing intervention to improve expectoration of airway secretions and prevent lung collapse in ventilated ICU patients: a randomized controlled trial. J Chin Med Assoc. 2009 Jun;72(6):316-22. doi: 10.1016/S1726-4901(09)70378-8. PMID 19541567